CLINICAL TRIAL: NCT06781814
Title: Research on the Role of Compound Probiotic Freeze-dried Powder in Improving Gastrointestinal Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WK20241231
Record Dates: First submitted 2025-01-01; First posted 2025-01-17 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Gastrointestinal Function
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wec600B group (Experimental): Participants will take the probiotic freeze-dried powder daily, each serving being 3.0 grams, to be consumed half an hour after meals.
  Interventions: Dietary Supplement: Probiotic
- Wec1000B group (Experimental): Participants will take the probiotic freeze-dried powder daily, each serving being 3.0 grams, to be consumed half an hour after meals.
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic — Probiotic strips with different strain formulas, specification: 3g/bag. Storage method: Keep away from light, seal tightly, and store in a cool, dry place.

SUMMARY:
This study aims to evaluate the effect of four high-activity compound probiotic freeze-dried powders on improving gastrointestinal function, observing their regulatory effects on the gut microbiota and the incidence of adverse reactions in study participants over a 4-week intervention period.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily, in writing, sign the informed consent form, agreeing to participate in this study
2. Able to complete the study according to the requirements of the trial protocol
3. Age between 18 and 65 years old
4. Meet the diagnostic criteria for gastrointestinal dysfunction established in the "Chinese Precision Health Communication Expert Consensus on Citizen's Guide to Gastrointestinal Health"
5. Symptoms: Irregular bowel movements, loose or hard stools, abdominal bloating, belching, flatulence, severe intestinal gas, abdominal pain, acid reflux, heartburn, pain in the stomach or abdomen when hungry, nausea
6. Signs: Abdominal pain and bloating, diarrhea and constipation, indigestion, gastric acid reflux, bad breath and foul-smelling flatulence, skin problems, changes in stool color and shape -

Exclusion Criteria:

1. Use of drugs affecting the intestinal flora (including antimicrobials, probiotics, intestinal mucosal protective agents, traditional Chinese patent medicines, etc.) for more than 1 week continuously within 1 month prior to screening
2. Short-term consumption of products similar to the test substance, which affects the judgment of the results
3. Use of antibiotics during illness
4. Participants with severe systemic diseases or malignant tumors
5. Participants allergic to any components of the compound probiotic freeze-dried powder used in this trial
6. Women who are pregnant or breastfeeding, or those who have plans to conceive in the near future
7. Participants who cannot participate in the trial due to personal reasons
8. Other participants deemed unsuitable for participation by the researcher -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-06-09 (Actual)

PRIMARY OUTCOMES:
Improvement of gastrointestinal function in study participants | 4 weeks
  Bowel movement frequency improvement: use the "bowel movement frequency scale" to record the number of bowel movements per week for participants, in order to assess changes in bowel movement frequency.

SECONDARY OUTCOMES:
Concentration of Short-Chain Fatty Acids in Fecal Samples | 4 weeks
  The concentration of short-chain fatty acids in fecal samples was determined by gas chromatography-mass spectrometry (GC-MS).
Metabolite Profile in Fecal Samples as an Indicator of Intestinal Microbiota Health | 4 weeks
  The metabolites in fecal samples were detected by liquid chromatography-mass spectrometry (LC-MS).

CONTACTS AND LOCATIONS:
Locations (1):
- School of Food and Bioengineering, Henan University of Science and Technology, Luoyang, Henan, China